CLINICAL TRIAL: NCT01639976
Title: Testing the Connection Between the Existence of Endometrial Flows With Doppler Examination if the Treatment Cytotec Success in Women With Miss Abortion
Brief Title: Doppler Flow Measurements in Patients With Misoprostol Treatment for Arrested Pregnancy
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hillel Yaffe Medical Center (Other Government)
Responsible Party: Sponsor
Other Study IDs: 0024-12
Record Dates: First submitted 2012-07-11; First posted 2012-07-13 (Estimated); Last update posted 2012-07-13 (Estimated); Status verified 2012-07

CONDITIONS: Missed Abortion
Keywords: Missed abortion, early pregnancy loss.
MeSH Terms: conditions — Abortion, Missed; Abortion, Spontaneous

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Testing the whether Doppler studies after cytotec treatment can predict success of treatment.

DETAILED DESCRIPTION:
All women who are treated with Cytotec for a missed abortion at 1st trimester will have a follow up ultrasound exam.

Doppler measurements will be performed but will be hidden from the clinicians. After the conclusion of treatment, data on Doppler would be vevealed in order to see if positive Doppler after Cytotec is predictive of failure of treatment or the need in several doses of cytotec.

ELIGIBILITY:
Inclusion Criteria:

* Women with miss abortion who choose treatment with cytotec

Exclusion Criteria:

Ages: 18 Years to 43 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Women with miss abortion who choose treatment with cytotec
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2012-09; Primary Completion 2013-09 (Estimated); Study Completion 2013-09 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Alon Shrim, MD, Principal Investigator — Hillel Yaffe Medical Center
Locations (1):
- Hillel Yaffe Medical Center, Hadera, Israel